CLINICAL TRIAL: NCT03106753
Title: Success of External Cephalic Version With Immediate Spinal Anesthesia Versus Spinal Anesthesia When Attempt Without Anesthesia Has Failed: A Randomized Controlled Trial
Brief Title: Success of External Cephalic Version Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis to assess concern for spinal anesthesia and increased cesarean delivery rate.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Natalie Porat, Resident, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-0236
Record Dates: First submitted 2017-03-27; First posted 2017-04-10 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: External Cephalic Version
Keywords: External Cephalic Version; neuraxial analgesia
MeSH Terms: interventions — Bupivacaine; Terbutaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spinal anesthesia immediately for ECV. (Active Comparator): The patient will have a spinal administered by the on call anesthesiologist using standard protocol (intrathecal bupivacaine 7.5 mg). The patient will then be administered 0.25 mg Terbutaline subcutaneously and the ECV will be attempted. Under ultrasound guidance the provider will attempt to lift the breech upward from the pelvis with one hand and guide the head with the other hand to produce a forward roll. If forward roll fails, a backward roll somersault may be attempted. ECV attempt will be abandoned if there is significant fetal bradycardia, discomfort to the patient, or if the procedure cannot be completed easily with these maneuvers. Once attempt is complete, whether successful or not, the patient will be monitored for a minimum of 30 minutes, and will be discharged once they are able to walk, void, and tolerate PO intake, only if fetal and maternal status is reassuring.
  Interventions: Drug: Bupivacaine; Drug: Terbutaline
- Spinal anesthesia if no intervention fails for ECV. (Experimental): The patient will be administered terbutaline 0.25 mg subcutaneously and the version will be attempted using the same procedure as above. If successful, the patient will be monitored for 30 minutes and discharged if fetal and maternal status is reassuring. If the attempt fails, the patient will be administered spinal anesthesia as above and the same maneuvers will be attempted. Once attempt is complete, whether successful or not, the patient will be monitored for a minimum of 30 minutes, and will be discharged once they are able to walk, void, and tolerate PO intake, only if fetal and maternal status is reassuring.
  Interventions: Drug: Bupivacaine; Drug: Terbutaline

INTERVENTIONS:
Drug: Bupivacaine — intrathecal bupivacaine 7.5 mg
Drug: Terbutaline — 0.25 mg Terbutaline subcutaneously

SUMMARY:
The purpose of this study is to determine the best way to optimize the success of external cephalic version (turning the baby from the outside). Attempting to turn babies in-utero is recommended because it may decrease the risk of needing a cesarean section for abnormal presentation. While the study team knows that this procedure can be effective, the study team still has some un-answered questions as to the best way to perform this procedure to increase the chance of success. Many prior studies have shown that using spinal anesthesia (a shot of medication placed in your back to numb and relax the abdomen) can increase the success rate of a version. This ultimately has led to the finding that using this anesthesia can decrease the rate of cesarean section. However, there have been only a small number of studies assessing the success rate if spinal anesthesia is used only in the event that without it fails. Therefore the study team is going to compare patients who receive spinal anesthesia with those who only receive spinal anesthesia if the procedure to turn the baby (ECV) fails without it.

DETAILED DESCRIPTION:
Breech presentation occurs in approximately 3-4% of term pregnancies and leads to one of the most common indications for cesarean delivery. Attempting an external cephalic version (ECV) significantly increases the chance of cephalic presentation at time of delivery and reduces the chance of cesarean section. Since ECV does in fact reduce the rate of cesarean section, many studies have sought to determine the best method to perform the procedure to optimize the chance of success. A recent meta-analysis concluded that administration of neuraxial analgesia significantly increases the success rate of ECV and also increases the incidence of vaginal delivery. However, there have been only 2 prospective studies and no randomized trials that evaluated the success of ECV using neuraxial analgesia only when initial attempt without it has failed. Therefore, the study team designed a randomized controlled trial with two groups: Group 1- patients receiving spinal anesthesia immediately versus Group 2- patients attempting ECV without spinal anesthesia with reattempt using a spinal if first attempt fails. This study will be conducted on labor and delivery at Mount Sinai West hospital. Patients who present to labor and delivery at term for ECV will be approached for enrollment and those who consent to be part of the study would be randomized into a group. ECV will then be attempted and delivery and neonatal outcomes will be collected. Patients will likely be enrolled in the study from time of version (approximately 37 weeks) until postpartum. This study will take approximately 1-2 years given the ECV rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients included are those with singleton pregnancies of at least 37 weeks gestation in nonvertex presentation with no contraindication for a vaginal delivery.
* Membranes must be intact with a minimum of a 2x2 pocket and Category 1 non-stress test.

Exclusion Criteria:

* All patients with a contraindication for a vaginal delivery will be excluded from the study.
* Patients with gross fetal anomalies or uterine malformations.
* Patients with contraindications to neuraxial anesthesia or allergies to any of the study medications will also be excluded.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Porat, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofmeyr GJ, Kulier R, West HM. External cephalic version for breech presentation at term. Cochrane Database Syst Rev. 2015 Apr 1;2015(4):CD000083. doi: 10.1002/14651858.CD000083.pub3. PMID 25828903
- [Background] Magro-Malosso ER, Saccone G, Di Tommaso M, Mele M, Berghella V. Neuraxial analgesia to increase the success rate of external cephalic version: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2016 Sep;215(3):276-86. doi: 10.1016/j.ajog.2016.04.036. Epub 2016 Apr 27. PMID 27131581
- [Background] Neiger R, Hennessy MD, Patel M. Reattempting failed external cephalic version under epidural anesthesia. Am J Obstet Gynecol. 1998 Nov;179(5):1136-9. doi: 10.1016/s0002-9378(98)70120-6. PMID 9822489
- [Background] Rozenberg P, Goffinet F, de Spirlet M, Durand-Zaleski I, Blanie P, Fisher C, Lang AC, Nisand I. External cephalic version with epidural anaesthesia after failure of a first trial with beta-mimetics. BJOG. 2000 Mar;107(3):406-10. doi: 10.1111/j.1471-0528.2000.tb13238.x. PMID 10740339

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Anesthesia Immediately for ECV.: The patient had a spinal administered by the on call anesthesiologist using standard protocol (intrathecal bupivacaine 7.5 mg). The patient was then administered 0.25 mg Terbutaline subcutaneously and the ECV was attempted. Under ultrasound guidance the provider attempt to lift the breech upward from the pelvis with one hand and guide the head with the other hand to produce a forward roll. If forward roll fails, a backward roll somersault may be attempted. ECV attempt will be abandoned if there is significant fetal bradycardia, discomfort to the patient, or if the procedure cannot be completed easily with these maneuvers. Once attempt is complete, whether successful or not, the patient will be monitored for a minimum of 30 minutes, and will be discharged once they are able to walk, void, and tolerate PO intake, only if fetal and maternal status is reassuring.
- Spinal Anesthesia if no Intervention Fails for ECV.: The patient was administered terbutaline 0.25 mg subcutaneously and the version was attempted using the same procedure. If successful, the patient was monitored for 30 minutes and discharged if fetal and maternal status is reassuring. If the attempt fails, the patient was administered spinal anesthesia and the same maneuvers attempted. Once attempt is complete, whether successful or not, the patient was monitored for a minimum of 30 minutes, and will be discharged once they are able to walk, void, and tolerate PO intake, only if fetal and maternal status is reassuring.
Period: Overall Study
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Started | 17 | 17
Completed | 17 | 16
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Spinal Anesthesia Immediately for ECV.: The patient had a spinal administered by the on call anesthesiologist using standard protocol (intrathecal bupivacaine 7.5 mg). The patient was then administered 0.25 mg Terbutaline subcutaneously and the ECV was attempted.
- Spinal Anesthesia if no Intervention Fails for ECV.: The patient was administered terbutaline 0.25 mg subcutaneously and the version was attempted. If the attempt fails, the patient was administered spinal anesthesia and the same maneuvers attempted. This group includes both those who did not require spinal anesthesia and those who subsequently require spinal anesthesia.
- Total: Total of all reporting groups
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV. | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (3.6) | 34.1 (4.6) | 33.7 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Parity [Count of Participants; unit: Participants] — The number of pregnancies reaching viable gestational age
  Participants
    0 | 13 | 13 | 26
    1 | 4 | 3 | 7
    2 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Success Rate of External Cephalic Version to Cephalic Presentation.
Description: Success rate will be measured by comparing the percentage of successful external cephalic versions in each group.
Time Frame: Day 1
Population: The data was analyzed by group, not by type of intervention (which means that for the delayed spinal group it was combined). This was done on purpose because the researchers wanted to compare the groups as a whole since that was what the researchers were looking at, the researchers were not comparing spinal versus no spinal.
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 17
Participants
  Nulliparous | 4 | 5
  Multiparous | 3 | 3

2. Secondary Outcome: Time From Procedure to Delivery.
Description: Number of days from procedure to delivery.
Time Frame: up to day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 17
hours | 12.6 (9.5) | 11.3 (7.7)

3. Secondary Outcome: Number of Participants With Various Mode of Delivery
Description: Mode of delivery as incidence of spontaneous vaginal delivery, operative vaginal delivery, or cesarean section.
Time Frame: up to day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 16
Participants
  Spontaneous Vaginal Delivery | 6 | 6
  Operative Vaginal Delivery | 0 | 1
  Cesarean Section | 11 | 9

4. Secondary Outcome: Numeric Rating Scale (NRS-11)
Description: Patient discomfort rated with NRS-11. Total scale from 0-10, with higher score indicating more pain.
Time Frame: Day 1
Population: Only those participants who underwent a second procedure completed the NRS-11 a second time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 17
score on a scale
  First procedure | 2.0 (2.3) | 6.1 (2.0)
  Second procedure: number analyzed (Participants) | 0 | 9
  Second procedure |  | 2.2 (2.9)

5. Secondary Outcome: Number of Adverse Events During Procedure
Description: Number of total specific adverse events such as: fetal bradycardia, emergent cesarean section, or abruption.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 17
events | 11 | 5

6. Secondary Outcome: Newborn Birth Weight
Description: Newborn birth weight in grams.
Time Frame: Day 1 of delivery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Spinal Anesthesia Immediately for ECV.: Newborn of the patients that had a spinal administered by the on call anesthesiologist using standard protocol (intrathecal bupivacaine 7.5 mg). The patient was then administered 0.25 mg Terbutaline subcutaneously and the ECV was attempted.
- Spinal Anesthesia if no Intervention Fails for ECV.: Newborns of the patient that was administered terbutaline 0.25 mg subcutaneously and the version was attempted. If the attempt fails, the patient was administered spinal anesthesia and the same maneuvers attempted. This group includes both those who did not require spinal anesthesia and those who subsequently require spinal anesthesia.
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 16
grams | 3321.6 (496.5) | 3257.7 (337.8)

7. Secondary Outcome: Number of Participants With Newborns With Apgar Score 7 or 9
Description: Newborns with Apgar Score 7 or 9 at 5 minutes after delivery. The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Time Frame: 7 minutes and 9 minutes after delivery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 16
Participants
  7 | 1 | 1
  9 | 16 | 15

8. Secondary Outcome: Cord pH
Description: Arterial cord pH level
Time Frame: Day 1
Population: Data results only for those who had arterial cord pH blood drawn,
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 8 | 7
pH | 7.2 (0.1) | 7.2 (0.1)

9. Secondary Outcome: Number of NICU Admission
Description: Number of patients whose neonate was admitted to the NICU in each group.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
Number analyzed (Participants) | 17 | 16
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 Day
Groups:
- Spinal Anesthesia Immediately for ECV.: The patient had a spinal administered by the on call anesthesiologist using standard protocol (intrathecal bupivacaine 7.5 mg). The patient was then administered 0.25 mg Terbutaline subcutaneously and the ECV was attempted.
  The data was analyzed by group, not by type of intervention (which means that for the delayed spinal group it was combined). This was done on purpose because the researchers wanted to compare the groups as a whole since that waa what the researchers were looking at, the researchers were not comparing spinal versus no spinal.
- Spinal Anesthesia if no Intervention Fails for ECV.: The patient was administered terbutaline 0.25 mg subcutaneously and the version was attempted. If the attempt fails, the patient was administered spinal anesthesia and the same maneuvers attempted. This group includes both those who did not require spinal anesthesia and those who subsequently require spinal anesthesia.
  The data was analyzed by group, not by type of intervention (which means that for the delayed spinal group it was combined). This was done on purpose because the researchers wanted to compare the groups as a whole since that waa what the researchers were looking at, the researchers were not comparing spinal versus no spinal.
Arm/Group | Spinal Anesthesia Immediately for ECV. | Spinal Anesthesia if no Intervention Fails for ECV.
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 11/17 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spinal Anesthesia Immediately for ECV. (N=17) | Spinal Anesthesia if no Intervention Fails for ECV. (N=17)
Bradycardia (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Nonreactive tracking (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Abruption (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cesarean Section (Pregnancy, puerperium and perinatal conditions) | 3 | 1
Hypotension (Cardiac disorders) | 7 | 2
Transient bradycardia (Pregnancy, puerperium and perinatal conditions) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03106753/Prot_SAP_000.pdf